CLINICAL TRIAL: NCT06609538
Title: The Impact of Preoperative Suggestions on Dreaming With Intravenous Sedation: A Randomized Controlled, Blinded Trial.
Brief Title: The Impact of Preoperative Suggestion on Dreaming
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wonkwang University Hospital (Other)
Responsible Party: Principal Investigator, Cheol Lee,MD,PhD,, Professor, M.D., Ph.D, Wonkwang University Hospital
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Wonkwang UH15
Record Dates: First submitted 2024-09-22; First posted 2024-09-24 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Dream, Day; Ketamine Adverse Reaction; Propofol Adverse Reaction
Keywords: Suggestion; dream incidence; dream contents; emotional tone; patient satisfaction
MeSH Terms: conditions — Patient Satisfaction | interventions — Control Groups; Propofol; Ketamine

STUDY DESIGN:
Intervention Model Description: 1. Control Group with Propofol: Receives standard preoperative instructions and propofol infusion.
  2. Suggestion Group with Propofol: Receives positive preoperative suggestions and propofol infusion.
  3. Control Group with Ketamine: Receives standard preoperative instructions and ketamine infusion.
  4. Suggestion Group with Ketamine: Receives positive preoperative suggestions and ketamine infusion.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Group with Propofol (Active Comparator): Receives standard preoperative instructions and propofol infusion.
  Interventions: Other: Control Group
- Suggestion Group with Propofol (Experimental): Receives positive preoperative suggestions and propofol infusion.
  Interventions: Other: Suggestion Group
- Control Group with Ketamine (Active Comparator): Receives standard preoperative instructions and ketamine infusion.
  Interventions: Other: Control Group
- Suggestion Group with Ketamine (Experimental): Receives positive preoperative suggestions and ketamine infusion.
  Interventions: Other: Suggestion Group

INTERVENTIONS:
Other: Control Group — Receives standard preoperative instructions and propofol or ketamine infusion.
  Other Names: Propofol; Ketamine
  Arms: Control Group with Ketamine; Control Group with Propofol
Other: Suggestion Group — Receives positive preoperative suggestions and propofol or ketamine infusion.
  Other Names: Propofol; Ketamine
  Arms: Suggestion Group with Ketamine; Suggestion Group with Propofol

SUMMARY:
Recent studies have shown that positive preoperative suggestions can significantly influence the quality of dreams and reduce the incidence of unpleasant dreams during sedation with agents like ketamine and propofol.

DETAILED DESCRIPTION:
Cheong et al. demonstrated that a simple positive suggestion before ketamine administration could reduce unpleasant dreams, while Kim et al. found that propofol, compared to midazolam, led to more vivid and memorable dreams, along with similar satisfaction levels in patients. This study aims to extend these findings by comparing the effects of propofol and ketamine sedation on dreaming during anesthesia, with a focus on how preoperative suggestions might influence dream content, emotional tone, and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 20-65 years.
* ASA physical status I-III.
* Scheduled for elective spinal anesthesia or brachial plexus block.
* Fluent in Korean.

Exclusion Criteria:

* Use of any medication, including premedication, within 12 hours before surgery.
* Cognitive impairments or psychiatric disorders (including a history of unpleasant dreams or nightmares).
* Current use of sedatives or hypnotics.
* History of severe or recurrent nightmares.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2024-09-19 (Actual); Primary Completion 2024-11-25 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Dreaming | Dreaming will be assessed immediately after full awakeness in the Post-Anesthesia Care Unit (PACU).
  The "Dreaming and Cognition Evaluation Questionnaire" will be used.questionnaire evaluates the incidence of dreaming, as well as the dream's content, emotional tone (rated on a 1-5 scale from very unpleasant to very pleasant), memorability, visual vividness, intensity, and other qualitative aspects such as sound, movement, and emotional significance.
Quality of Dreaming | Dreaming will be assessed immediately in the Post-Anesthesia Care Unit (PACU).
  The "Dreaming and Cognition Evaluation Questionnaire" will be used. This questionnaire evaluates the incidence of dreaming, as well as the dream's content, emotional tone (rated on a 1-5 scale from very unpleasant to very pleasant), memorability, visual vividness, intensity, and other qualitative aspects such as sound, movement, and emotional significance.

SECONDARY OUTCOMES:
Satisfaction with Care | Satisfaction will be assessed immediately after full awakeness in the Post-Anesthesia Care Unit (PACU)
  A 101-point numerical rating scale included in the "Dreaming and Cognition Evaluation Questionnaire" will be used to measure patient satisfaction with the overall care and sedation experience.
Adverse events | Monitoring will be continuous with regular vital signs recorded every 5 minutes during surgery and every 15 minutes in the PACU.
  Any complications such as hypotension,or bradycardia, will be recorded systematically.

CONTACTS AND LOCATIONS:
Overall Officials: Cheol Lee, M.D.,Ph.D, Study Director — Wonkwang University Hospital
Locations (1):
- WonwangUH, Iksan, Please Select, South Korea